CLINICAL TRIAL: NCT02488681
Title: Medtronic Micra Transcatheter Pacing System Continued Access Study
Brief Title: Micra Transcatheter Pacing System Continued Access Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Micra CA
Record Dates: First submitted 2015-06-18; First posted 2015-07-02 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micra Pacemaker Implant (Experimental): Micra Pacemaker Implant
  Interventions: Device: Micra Pacemaker Implant

INTERVENTIONS:
Device: Micra Pacemaker Implant

SUMMARY:
Medtronic is sponsoring the Micra Continued Access (CA) study to provide continued access to the Micra System while the marketing application is under review by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The Micra CA study is a prospective, non-randomized, multi-center, study designed to allow controlled access of the Micra system when used as intended. All subjects enrolled in the Micra CA Study will be prospectively followed from implant, at 6-month intervals until study closure (i.e. FDA approval). Patients with previous or existing inactive implanted cardiac stimulation systems will have additional follow ups.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Subject meets Class I or ll indication for implantation of single chamber ventricular pacemaker and is intended to be implanted with a Micra System
* Subject able and accessible for follow-up per study requirements
* Subject is at least 18 years of age
* Patient is not enrolled in a concurrent drug and/or device study that may confound registry result.

Exclusion Criteria:

* Subject has had an acute myocardial infraction (AMI) within 30 days of implant
* Subject has implantation of neurostimulator or any other chronically implanted device which uses current in the body
* Subject with mechanical tricuspid valve, implanted vena cava filter, or left ventricular assist device (LVAD)
* Subjects who are morbidly obese and physician believes telemetry communication of ≤5 inches (12.5 cm) could not be obtained with programmer head.
* Subject who femoral venous anatomy is unable to accommodate a 23 French introducer sheath or implant on the right side of the heart (for example due to obstructions or sever tortuosity) in the opinion of the implanter
* Subjects with known intolerance to Nickel-Titanium (Nitinol) Alloy
* Subject for whom a single dose of 1.0mg dexamethasone acetate may be contraindicated
* Subjects with life expectancy less than 12-months
* Subject is enrolled in a concurrent drug and/or device study that may confound CA study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Baptist Heart Specialists, Jacksonville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Iowa Heart Center, West Des Moines, Iowa
  - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Mid America Heart Institute, Kansas City, Missouri
  - Morristown Memorial Hospital, Morristown, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - North Shore LIJ Health System, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - Providence Health and Services, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Vanderbilt University Medical Center Heart and Vascular Institute, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - CHI Saint Luke's Health - Baylor Saint Luke's Medical Center, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Piccini JP, Cunnane R, Steffel J, El-Chami MF, Reynolds D, Roberts PR, Soejima K, Steinwender C, Garweg C, Chinitz L, Ellis CR, Stromberg K, Fagan DH, Mont L. Development and validation of a risk score for predicting pericardial effusion in patients undergoing leadless pacemaker implantation: experience with the Micra transcatheter pacemaker. Europace. 2022 Jul 21;24(7):1119-1126. doi: 10.1093/europace/euab315. PMID 35025987
- [Derived] El-Chami MF, Shinn T, Bansal S, Martinez-Sande JL, Clementy N, Augostini R, Ravindran B, Sagi V, Ramanna H, Garweg C, Roberts PR, Soejima K, Stromberg K, Fagan DH, Zuniga N, Piccini JP. Leadless pacemaker implant with concomitant atrioventricular node ablation: Experience with the Micra transcatheter pacemaker. J Cardiovasc Electrophysiol. 2021 Mar;32(3):832-841. doi: 10.1111/jce.14881. Epub 2021 Jan 23. PMID 33428248
- [Derived] Garg A, Koneru JN, Fagan DH, Stromberg K, Padala SK, El-Chami MF, Roberts PR, Piccini JP, Cheng A, Ellenbogen KA. Morbidity and mortality in patients precluded for transvenous pacemaker implantation: Experience with a leadless pacemaker. Heart Rhythm. 2020 Dec;17(12):2056-2063. doi: 10.1016/j.hrthm.2020.07.035. Epub 2020 Aug 4. PMID 32763431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 285 subjects were consented at 31 research centers in the United States from June 2015 to April 2016 when FDA approval was obtained.
Pre-assignment Details: Of the 285 patients that were consented to participate in the study, 276 patients underwent a Micra implant attempt. Nine patients who were consented into the study did not ultimately have a Micra implant attempt prior to study closure.
Groups:
- Micra Pacemaker Implant: Patients who underwent a Micra implant attempt
Period: Overall Study
Arm/Group | Micra Pacemaker Implant
Started | 276 (Patients with Micra implant attempt)
Completed | 269 (Patients successfully implanted with Micra)
Not Completed | 7
Not completed — Implant unsuccessful | 7

BASELINE CHARACTERISTICS:
Population: Patients with a Micra implant attempt
Groups:
- Micra Pacemaker Implant: All subjects who attempted Micra implant procedure
Arm/Group | Micra Pacemaker Implant
Number analyzed (Participants) | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121
  Male | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 264
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 248
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 276

OUTCOME MEASURES:

1. Primary Outcome: Complications
Description: Micra system and/or procedure-related complication rate
Time Frame: 3 months post last follow up
Population: All subjects who attempted Micra implant procedure
Measure: Number (95% Confidence Interval); unit: % participants with complication
Arm/Group | Micra Pacemaker Implant
Number analyzed (Participants) | 276
% participants with complication | 4 [2 to 7]

ADVERSE EVENTS:
Time Frame: From implant attempt to last subject follow-up, ranging from 0 to approximately 12 months.
Arm/Group | Micra Pacemaker Implant
Serious Adverse Events (participants affected / at risk) | 27/276
Other Adverse Events (participants affected / at risk) | 16/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micra Pacemaker Implant (N=276)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Cardiac perforation (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Device capturing issue (General disorders) | 1 (2)
Device pacing issue (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micra Pacemaker Implant (N=276)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Cardiac discomfort (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Device capturing issue (General disorders) | 1 (1)
Device pacing issue (General disorders) | 4 (4)
Incision site infection (Infections and infestations) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 3 (3)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and Participating Institutions will provide any publication of Study Data generated by PI and/or Participating Institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.